CLINICAL TRIAL: NCT03229031
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 3 Study to Evaluate the Safety and Efficacy of ES135 in Subjects With Spinal Cord Injury
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: low recruitment rate
Sponsor: Eusol Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ES135-1601
Record Dates: First submitted 2017-07-20; First posted 2017-07-25 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord, spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomized, Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ES135 (Experimental)
  Interventions: Drug: ES135
- Placebo (Placebo Comparator)
  Interventions: Drug: ES135

INTERVENTIONS:
Drug: ES135 — ES135 will be administered via intrathecal

SUMMARY:
To demonstrate the superior effect of ES135 combined with spinal cord repairing surgery, compared to a placebo control with spinal cord repairing surgery, on post-surgery motor function recovery as measured by the changes from baseline of ISNCSCI Motor Scores in subjects

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of either sex and 15-65 years of age.
2. Subjects have spinal cord injury and the subjects must be categorized as Grade A or B by the ASIA Impairment Scale.
3. Subjects have adequate heart, lung, kidney and liver function.
4. Subjects are able to give voluntary and dated informed consent prior to enrollment.

Exclusion Criteria

1. Penetration SCI
2. Brain damage or multiple injuries
3. History of congenital or acquired abnormalities in the spinal cavity
4. History of congenital or acquired immunodeficiency disorders
5. History of malignancies or positive results
6. Current serious/uncontrollable infections or others serious diseases
7. Pregnant or lactating women
8. Allergy to ES135 or any of its excipients
9. Unable to obtain informed consent from subject

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-03-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change of International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Motor Scores | 48 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Taipei Veterans General Hospital, Taipei